CLINICAL TRIAL: NCT03904862
Title: PBTC-053: A Pediatric Brain Tumor Consortium Phase I/ II and Surgical Study of CX-4945 in Patients With Recurrent SHH Medulloblastoma
Brief Title: Testing the Safety and Tolerability of CX-4945 in Patients With Recurrent Medulloblastoma Who May or May Not Have Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The decision to permanently close PBTC-053 was made following communication from the NCI that the PBTC grant will not be extended beyond March 31, 2026.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: Senhwa Biosciences, Inc. (Industry); National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-053; UM1CA081457 (NIH); NCI-2019-00180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-053 (Other: Pediatric Brain Tumor Consortium); PBTC-053 (Other: CTEP)
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Medulloblastoma, Childhood; Medulloblastoma Recurrent; Medulloblastoma
Keywords: Medulloblastoma; Sonic Hedgehog (SHH) positive
MeSH Terms: conditions — Medulloblastoma; Microphthalmia, Isolated, with Coloboma 5 | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Skeletally-immature (Experimental): Skeletally-immature children with refractory or recurrent medulloblastoma of the SHH group
  Interventions: Drug: CX 4945
- Phase II - Skeletally-mature (Experimental): Skeletally-mature subjects with refractory or recurrent medulloblastoma of the SHH group
  Interventions: Drug: CX 4945
- Surgical (Experimental): Subjects who are eligible for the Phase I or Phase II arm of the trial and are candidates for surgery, may be enrolled in the surgical arm prior to initiation of the Phase I or Phase II treatment.
  Interventions: Drug: CX 4945

INTERVENTIONS:
Drug: CX 4945 — CX-4945 is supplied as 200 mg capsules delivered orally as a formulated API
  Other Names: Silmitasertib sodium

SUMMARY:
This is a multi center, Phase I, Phase II and surgical study of the CX-4945 drug (silmitasertib sodium) for patients with recurrent SHH (Sonic Hedgehog) medulloblastoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and recommend a Phase II dose of CX-4945 administered orally daily to skeletally-immature children with recurrent SHH (sonic hedgehog) medulloblastoma (Phase I) II. To describe the toxicity profile and define the dose-limiting toxicities associated with CX-4945 in children with recurrent SHH (Sonic hedgehog) medulloblastoma (Phase I) III. To characterize the pharmacokinetics of CX-4945 administered on this schedule in skeletally-immature children with recurrent SHH medulloblastoma (Phase I) IV. To characterize the concentrations of CX-4945 in tumor after administration of CX-4945 and surgical resection (Surgical Study). V. To establish the safety and characterize the toxicity of 1000mg BID continuous dosing of CX-4945 in skeletally-mature patients with recurrent SHH medulloblastoma (Phase II). VI. To estimate the objective response rate associated with CX-4945 in skeletally-mature patients with recurrent SHH medulloblastoma

SECONDARY OBJECTIVES:

I. To document preliminary antitumor activity of CX-4945 in skeletally-immature children with recurrent SHH medulloblastoma (Phase I). II. To perform a genomic analysis within the confines of a Phase I study to investigate correlation between response to treatment and the presence of specific genomic alterations. and/or specific subgroups of disease (Phase I). III. To explore the ability of CX-4945 at the MTD/ RP2D to inhibit CK2-mediated signaling in tumor (Surgical Study). IV. To characterize the pharmacokinetics of CX-4945 in skeletally-mature patients with recurrent SHH medulloblastoma (Phase II). V. To perform a genomic analysis within the confines of a Phase II study to investigate correlation between response to treatment and the presence of specific genomic alterations and/or specific subgroups of disease (Phase II).

OUTLINE: Phase I component is a dose-escalation study. The Phase II component is to establish the safety of 1000mg BID given continuously.

The study will open with a safety cohort of 3 subjects who are considered skeletally-mature. The initial 3 subjects will be administered CX-4945 twice a day at the adult RP2D of 1000 mg BID or at its BSA adjusted equivalent; however, the dose will be given continuously. If there are not excessive toxicities in this cohort, the study will proceed following the Phase II design for subjects who are skeletally-mature.

Following the safety lead in, the Phase 1 component of this trial will be initiated. Skeletally-immature children with refractory or recurrent medulloblastoma of the SHH subgroup, will be administered CX-4945 twice a day on a continuous basis at a starting dose of 600mg/m2 BID which corresponds approximately to the BSA adjusted recommended Phase 2 dose (RP2D) of 1000mg. The Phase 1 study will escalate doses to determine the maximum tolerated dose skeletally-immature children.

The surgical study will be initiated after the first 3 patients in the skeletally-mature cohort are treated for initial assessment of safety and did not experience excessive toxicity. Skeletally-mature subjects with recurrent or refractory SHH medulloblastoma will be eligible as soon the surgical study is initiated and will receive drug at 1000mg BID or its BSA adjusted equivalent depending upon age and BSA. Skeletally-immature subjects will only be eligible to enroll on the surgical trial once the MTD is defined in the Phase 1 component and will receive drug at the established MTD for this cohort.

After completion of study treatment, patients are followed up to 2 years.

ELIGIBILITY:
Screening Criteria:

1. Tumor

   a. Patient must have a diagnosis of medulloblastoma that is recurrent or progressive. All tumors must have histologic verification either at the time of diagnosis or recurrence.
2. Adequate Pre-trial Tumor Tissue a. Patient must have adequate pre-trial tumor material available for subgrouping.
3. Prior Therapy

   a. Patient must have received and failed standard therapy for medulloblastoma.
4. Screening Consent a. Participant is willing to sign a screening consent. The screening consent is for subgroup testing for all participants and for bone age determination in subjects ≤ 18 years. The screening consent is to be obtained according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.

Inclusion Criteria:

1. Phase I Skeletally-immature:

   1. Patient must be skeletally-immature at the time of study enrollment, defined as females with a bone age < 14 years and males with a bone age < 16 years.
   2. Patients who participate in the expansion cohort must have bi-dimensionally measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions (Section 12.2.2). Patients with measurable extraneural disease only are also eligible.
   3. Patient must be ≥ 3 and ≤ 18 years of age at the time of enrollment.
   4. Patients enrolled on the Phase I study must have a BSA as noted below:

   Dose Level 0 (400 mg/m2 BID): Minimum - 0.84m2; Maximum - 2.25m2 Dose Level 1 (600 mg/m2 BID): Minimum - 0.60m2; Maximum - 2.00m2 Dose Level 2 (800 mg/m2 BID): Minimum - 0.63m2; Maximum - 2.00m2
2. Phase II Skeletally-mature:

   a. Patients must be skeletally-mature, defined as females with a bone age ≥14 years and males with a bone age ≥ 16 years OR have a chronological age >18 years.

   b. Patients must have bi-dimensionally measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions. Patients with measurable extraneural disease only are also eligible.
3. Surgical Study:

   1. Surgical resection must be clinically indicated.
   2. Must be ≥3 years at time of enrollment.
   3. Must be amenable to receiving CX-4945 for 5-7 days prior to surgery
4. All Phases:

   1. Patient must have a diagnosis of SHH medulloblastoma that is recurrent or progressive, confirmed histologically and by CLIA-certified methylation-based subgroup testing at Cincinnati Children's Hospital Medical Center (CCHMC), Memorial Sloan Kettering Cancer Center (MSKCC), National Cancer Institute (NCI), or Nationwide Children's Hospital (NCH). Results from prior testing at these designated sites using the same approaches described for this study will be accepted.
   2. Prior Therapy

      • Must have received prior therapy which included radiation therapy and recovered from acute treatment related toxicities.

      • Must have received the last dose of myelosuppressive therapy at least 21 days prior to enrollment and at least 42 days if nitrosourea.

      • Must have received the last dose of another investigational or biologic agent ≥7 days prior. For agents known to have adverse events occurring beyond 7 days, the period must be extended to accommodate the longer interval. For monoclonal antibodies with prolonged half-lives, at least 3 half-lives must have elapsed.

      • Must have received last fraction of craniospinal or total body irradiation or radiation to ≥50% of the pelvis >12 weeks prior to enrollment. Last fraction of focal irradiation must be >4 weeks prior to enrollment.

      • Must be ≥ 24 weeks since allogeneic stem cell transplant with no evidence of acute graft vs. host disease.

      • Must be ≥12 weeks since autologous stem cell transplant.
   3. Must be off all colony-forming growth factors at least 1 week prior to enrollment. Must be off 2 weeks if the subject received a long-acting formulation.
   4. If neurological deficits are present, must have been stable for a minimum of 1 week prior to enrollment.

      • Patients with seizure disorders may be enrolled if seizures are well controlled.
   5. Must have a Karnofsky/Lansky Performance status ≥50%
   6. Must have adequate organ and marrow function
   7. Subjects receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment.
   8. Female patients of childbearing potential must have a negative pregnancy test.
   9. Patients of child-bearing or child fathering potential must be willing to use medically acceptable form of birth control while treated on this study and for 3 months after drug cessation.
   10. Parent or legal guardian must be able to understand and willing to sign the written informed consent.

C. Exclusion Criteria:

1. All Phases

1. Nursing mothers due to an unknown but potential risk for adverse events in nursing infants.
2. Patients with a history of any other malignancy with the exception of patients with a secondary brain tumor if the patient's prior malignancy has been in remission for at least 5 years from the end of treatment.
3. Patients with any of the following gastrointestinal disorders - difficulty swallowing or active malabsorption, uncontrolled diarrhea, gastritis, ulcerative colitis, Crohn's disease or hemorrhagic coloproctitis, history of gastric or small bowel surgery involving any extent of gastric or small bowel resection.
4. Patients with any clinically significant unrelated systemic illness that would compromise the patient's ability to tolerate therapy, put them at additional risk for toxicity or interfere with the study procedures or results.
5. Corrected QT (QTc) interval is >480ms
6. Patients who are receiving other anti-cancer or investigational drug therapy
7. Patients who are on warfarin or statins.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose of CX-4945 | 4 weeks
  Defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic.
Phase I: Plasma pharmacokinetics of CX-4945 in skeletally-immature children | 4 weeks
  To report the plasma drug concentration of CX-4945 on this schedule in skeletally-immature children
Surgical Study: Intratumoral PK concentrations | Prior to starting CX-4945 (Day -5 or -7), prior to dose on Day -3, prior to dose on Day -1, day of surgery and during surgery at the time of tissue collection
  Average tumor CX-4945 concentrations.
Phase II: Sustained objective response rate (PR-CR) rate in the skeletally mature cohort | Up to 2 years from enrollment
  Percentage of patients who achieve sustained objective response.

SECONDARY OUTCOMES:
Progression free survival | Up to 3 years from enrollment
  Interval of time between the date of initiation of protocol treatment and minimum date of documentation of PD, second malignancy, death due to any cause or date of last follow-up.
Objective response rate in the skeletally-immature cohort | Up to 2 years from enrollment
  Percentage of patients who achieve objective response in the skeletally-immature cohort
Plasma pharmacokinetics of CX-4945 in skeletally-mature subjects | 4 weeks
  To report the plasma drug concentration of CX-4945 in skeletally-mature subjects
Relative frequency of genomic alterations in archival tissue | At time of enrollment
  Percentage of various genomic alterations will be reported
Surgical study: Reduction in CK2-mediated signaling in tumor. | 4 weeks
  Change in CK2 activity in tumor tissue from patients on the surgical are at baseline and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Salloum, MD, Study Chair — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University and Lucile Packard Children's Hospital, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas